CLINICAL TRIAL: NCT06173531
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Parallel-group Study of Carbetocin Nasal Spray for the Treatment of Hyperphagia in Prader-Willi Syndrome
Brief Title: Study of Carbetocin Nasal Spray for the Treatment of Hyperphagia in Prader-Willi Syndrome
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACP-101-302; 2023-506200-24-00 (EU CTIS Number)
Record Dates: First submitted 2023-12-08; First posted 2023-12-15 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Hyperphagia in Prader-Willi Syndrome
Keywords: Randomized; Placebo-controlled
MeSH Terms: interventions — carbetocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Carbetocin (Experimental): Carbetocin nasal spray 3.2 mg three times daily (TID)
  Interventions: Drug: Carbetocin
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Carbetocin — Carbetocin nasal spray 3.2 mg three times daily (TID)
  Other Names: ACP-101
  Arms: Carbetocin
Drug: Placebo — Placebo given TID, identical in appearance respective to carbetocin treatment
  Arms: Placebo

SUMMARY:
12-week, randomized, double-blind, placebo-controlled, parallel-group study of carbetocin nasal spray for the treatment of hyperphagia in Prader-Willi syndrome (PWS)

DETAILED DESCRIPTION:
This is a 12-week, multicenter, randomized, double-blind, placebo-controlled, parallel-group study comparing carbetocin nasal spray 3.2 mg TID with placebo (matched placebo nasal spray TID) in subjects with PWS.

ELIGIBILITY:
Inclusion Criteria

* Male or female and 5 through 30 years of age
* Prader-Willi syndrome with a documented disease-causing mutation
* Increased appetite with decreased satiety accompanied by food seeking (consistent with PWS Nutritional Phase 3)
* HQ-CT total score of ≥13 at Screening and Baseline
* CGI-S score for hyperphagia in PWS of ≥4 at Screening and Baseline
* Lives with a caregiver who understands and is willing and able to adhere to study-related procedures and is willing to participate in all study visits

Exclusion Criteria

* Genetically diagnosed with Schaaf-Yang syndrome or another genetic, hormonal, or chromosomal cognitive impairment besides PWS
* An active upper respiratory infection at the Screening visit or the Baseline visit
* Any clinically significant cardiovascular disorder, renal, hepatic, gastrointestinal, or respiratory disease, including severe asthma
* History of, or current, cerebrovascular disease, brain trauma, epilepsy, or frequent migraines. A history of febrile seizures is not exclusionary
* Nasal surgery within 1 month of Screening visit or planning to have nasal surgery during the study.
* Unwilling to abstain from nasal saline, other nasal irrigation, and other intranasal medications during the Screening period and through the treatment period of the study
* Clinically significant irritability or agitation, requiring initiation of or increase in the dose of antipsychotic medication, within the 6 months prior to the Screening visit
* Used prostaglandins, prostaglandin analogues, or prostaglandin agonists in the 3 months prior to the Baseline visit. Inhibitors of prostaglandin synthesis, such as nonsteroidal anti-inflammatory drugs, are not exclusionary.
* Started a glucagon-like peptide 1 (GLP-1) agonist within the 6 months prior to the Screening visit. Treatment with GLP-1 agonist is allowed if the subject has been taking it for more than 6 months prior to Screening.
* Used oxytocin, desmopressin (DDAVP), tesofensine, diazoxide choline, melanocortin-4 receptor (MC4R) agonists (e.g., setmelanotide), or any medication approved to treat hyperphagia within 6 months prior to the Baseline visit
* Active psychotic symptoms, a history of psychotic symptoms, or a psychotic disorder
* History of suicide attempt or inpatient psychiatric hospitalization
* New food-related interventions, including environment or dietary restrictions, within 1 month prior to the Screening visit or during the Screening period (i.e., before the Baseline visit)

Additional inclusion/exclusion criteria apply. Subjects will be evaluated at screening to ensure that all criteria for study participation are met.

Ages: 5 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 170 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline at Week 12 in caregiver-rated Hyperphagia Questionnaire for Clinical Trials (HQ-CT) score | Baseline to Week 12
  The HQ-CT is a nine-item questionnaire designed to be completed by caregivers of subjects with PWS. It is a revision of the 11-item HPWSQ-R and has been further validated. The Foundation for Prader-Willi Research has made the HQ-CT available for clinical studies in PWS, and it is the consensus instrument within the PWS research community for measuring observable behaviors that stem from subjects' excessive drive to eat.
  The HQ-CT should be completed by the same caregiver throughout the study. The HQ-CT will be administered to the caregiver by a rater using standardized prompts. The Food Safe Zone should be administered immediately before administration of the HQ-CT.
  A higher score on the HQ-CT indicates greater severity of hyperphagia.

SECONDARY OUTCOMES:
Change from Baseline at Week 12 in caregiver-rated Clinical Global Impression-Severity (CGI-S) score for PWS | Baseline to Week 12
  The CGI-S is a rating scale that records a clinician's global impression of the current severity of illness on a seven-point scale, using a range of responses from 1 (normal) to 7 (among the most severely ill subjects).
Clinical Global Impression-Change (CGI-C) for PWS score at Week 12 | Score at Week 12
  The CGI-C is a rating scale that records a clinician's global impression of change in severity of illness, using a range of responses from 1 (very much improved) to 7 (very much worse).

CONTACTS AND LOCATIONS:
Locations (30):
- United States (19):
  - Children's of Alabama, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - University of California Irvine, Orange, California
  - Stanford University School of Medicine, Palo Alto, California
  - Rady Children's Hospital San Diego, San Diego, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Mercy Hospital, Kansas City, Missouri
  - SSM Health/Saint Louis University, St Louis, Missouri
  - Maimonides Medical Center, Brooklyn, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - UPMC-Children's Hospital Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt Clinical Research Center, Nashville, Tennessee
  - Cook Children's Health Care System, Fort Worth, Texas
  - Christus Children's, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- Canada (2):
  - Alberta Diabetes Institute, Edmonton, Alberta
  - CHU Sainte Justine, Montreal, Quebec
- Centre Hospitalier Universitaire (CHU) de Toulouse - Hôpital des Enfants, Toulouse, France
- Germany (2):
  - KJF Klinik Josefinum gGmbH, Augsburg
  - Universitätsklinikum Essen, Essen
- Spain (3):
  - Parc Taulí Hospital Universitari, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
- United Kingdom (3):
  - University Hospitals Birmingham NHS Foundation Trust - Heartlands Hospital, Birmingham
  - Royal Hospital for Children Glasgow Clinical Research Facility, Glasgow
  - Barts Health NHS Trust - The Royal London Hospital, London

IPD SHARING:
Plan to Share IPD: No